CLINICAL TRIAL: NCT01354366
Title: The Effects on Growth and Tolerance of Hypoallergenic Formulas Fed to Term Infants
Brief Title: Growth and Tolerance of Hypoallergenic Formulas
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Timothy Cooper, M.D., Mead Johnson Nutrition
Other Study IDs: 3383-1
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Growth of Term Infants
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Marketed hypoallergenic infant formula containing a probiotic
  Interventions: Other: Infant formula
- Experimental 1: An investigational hypoallergenic infant formula with a different protein content, containing the same probiotic as the control
  Interventions: Other: Infant formula
- Experimental 2: An investigational hypoallergenic infant formula with a different protein content, without a probiotic
  Interventions: Other: Infant formula

INTERVENTIONS:
Other: Infant formula

SUMMARY:
This clinical trial will evaluate two investigational hypoallergenic infant formulas with a differing protein content to determine if they provide normal growth and are well tolerated by term infants as compared to a marketed hypoallergenic formula.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 12-16 days of age at randomization
* Term infant with birth weight of a minimum of 2500 grams
* Solely formula fed
* Signed Informed Consent and Protected Health Information

Exclusion Criteria:

* History of underlying metabolic or chronic disease or immunocompromised
* Feeding difficulties or formula intolerance

Ages: 12 Days to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Heatly, term infants
Sampling Method: Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Body weight measured at each study visit | 3.5 months

SECONDARY OUTCOMES:
Recall of infant formula intake at each study visit | 3.5 months
Body Length and Head Circumference measured at each study visit | 3.5 months
Recall of stool characteristics and tolerance at each study visit | 3.5 months
Medically-confirmed adverse events collected throughout the study period | 3.5 months
Parental Product Assessment Questionnaire completed at Study Visit 2 | once

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cooper, M.D., Study Director — Mead Johnson Nutrition
Locations (24):
- United States (24):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Pediatrics East - Alabama Clinical Therapeutics, Pinson, Alabama
  - Central Arkansas Pediatric Clinic, Benton, Arkansas
  - The Children's Clinic of Jonesboro, Jonesboro, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Norwich Pediatric Group, P.C., Norwich, Connecticut
  - Altamonte Pediatric Associates, Lake Mary, Florida
  - Children's Medical Association, Plantation, Florida
  - North Georgia Clinical Research Center/White's Pediatrics, Dalton, Georgia
  - Deaconess Clinic, Newburgh, Indiana
  - PTCU/Children and Youth Project, Louisville, Kentucky
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Woburn Pediatric Associates, Woburn, Massachusetts
  - Gretchen Swanson Center for Nutrition, Omaha, Nebraska
  - Capital Pediatrics & Adolescent Center, Raleigh, North Carolina
  - Innovis Health South University, Fargo, North Dakota
  - Pediatric Associates of Mt. Carmel, Inc, Cincinnati, Ohio
  - Pediatric Associates of Fairfield, Inc, Fairfield, Ohio
  - Red Lion Pediatrics, Philadelphia, Pennsylvania
  - Primary Physicians Research, Inc, Pittsburgh, Pennsylvania
  - The Jackson Clinic - North Jackson, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Austin Diagnostic Clinic, Austin, Texas

REFERENCES:
- [Derived] Adams CB, Johnston WH, Deulofeut H, Leader J, Rhodes R, Yeiser M, Harris CL, Wampler JL, Hill RJ, Cooper T. Growth and tolerance of healthy, term infants fed lower protein extensively hydrolyzed or amino acid-based formula: double-blind, randomized, controlled trial. BMC Pediatr. 2021 Jul 21;21(1):323. doi: 10.1186/s12887-021-02617-z. PMID 34289820